CLINICAL TRIAL: NCT00219011
Title: A Twelve-week, Randomized, Double-blind, Multi-center, Placebo Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of Aliskiren 150 mg When Added to Standard Therapy in Hypertensive Patients With Stable Heart Failure
Brief Title: "ALOFT - Aliskiren Observation of Heart Failure Treatment": Efficacy and Safety of Aliskiren Added on Top of Standard Therapy in Adults (≥ 18 Years) With Stable Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CSPP100A2313
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure
Keywords: Aliskiren, heart failure,hypertension
MeSH Terms: conditions — Heart Failure; Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
This study was designed to determine if patients, who have both high blood pressure and heart failure and are currently receiving drug treatment for heart failure, have an improvement in their heart failure signs and symptoms and other indicators of heart failure after being treated with aliskiren on top of their current heart failure treatment. Aliskiren is an investigational drug; its safety will also be evaluated in this trial.

ELIGIBILITY:
Inclusion Criteria:

* History of diagnosis or currently have high blood pressure
* Stable heart failure (NYHA Class 2-4) for at least 1 month before study entry. Subject should be on a stable dose regimen of heart failure medication.
* Brain natriuretic peptide (BNP) > 150 pg/ml at baseline (to be evaluated by physician at first visit)

Exclusion Criteria:

* Previous treatment with aliskiren
* High blood pressure due to secondary reasons or constant low blood pressure (systolic < 90 mmHg)
* History of heart attack or coronary bypass surgery in the past 6 months

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2005-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Measurement of safety information and tolerability of drug after 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the heart failure biochemical markers of N-terminal pro-brain natriuretic peptide (NT-proBNP) and brain natriuretic (BNP) after 12 weeks
Change from baseline in aldosterone (a steroid hormone secreted by the adrenal cortex that regulates salt and water balance in the body) after 12 weeks
Changes in New York Heart Association heart failure stages after 12 weeks
Changes from baseline in the forces of the circulation of blood as measured by echocardiography to after 12 weeks
Change from baseline in mean sitting systolic and diastolic blood pressure after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Jackson CE, MacDonald MR, Petrie MC, Solomon SD, Pitt B, Latini R, Maggioni AP, Smith BA, Prescott MF, Lewsey J, McMurray JJ; ALiskiren Observation of heart Failure Treatment (ALOFT) investigators. Associations of albuminuria in patients with chronic heart failure: findings in the ALiskiren Observation of heart Failure Treatment study. Eur J Heart Fail. 2011 Jul;13(7):746-54. doi: 10.1093/eurjhf/hfr031. Epub 2011 Apr 1. PMID 21459891
- [Derived] McMurray JJ, Pitt B, Latini R, Maggioni AP, Solomon SD, Keefe DL, Ford J, Verma A, Lewsey J; Aliskiren Observation of Heart Failure Treatment (ALOFT) Investigators. Effects of the oral direct renin inhibitor aliskiren in patients with symptomatic heart failure. Circ Heart Fail. 2008 May;1(1):17-24. doi: 10.1161/CIRCHEARTFAILURE.107.740704. PMID 19808266